CLINICAL TRIAL: NCT04579432
Title: The Effect of Web Based Reproductive Health Education on Sexual Myths and Risky Behaviors in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Güzin Ünlü, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 58797649-050-
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Health Risk Behaviors; Reproductive Health; Sexual Health
Keywords: Health Risk Behaviors; Reproductive Health; Sexual Health; Sexual Myths
MeSH Terms: conditions — Health Risk Behaviors | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: There is a control group and an experimental group in this research. Pre-test and post-test will be carried out with a pattern. A pre-test will be made to the control and experimental groups simultaneously. Then, the experimental group will be trained and the final test will be conducted simultaneously with the non-intervened control group.
Who Masked: Participant
Masking Description: The participants will not know which group they are in. they won't interact with each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental)
  Interventions: Other: Education
- Control Group (No Intervention)

INTERVENTIONS:
Other: Education — With the training module prepared according to the ADDIE model, the intervention group will be trained on reproductive health and sexual health.
  Arms: Training Group

SUMMARY:
The World Health Organization (WHO) defines the concept of reproductive health as "not only the absence of disease or disability, but a state of complete physical, mental and social welfare in all matters related to the reproductive system, functions and processes". However, it also emphasizes that people have free will in the timing of having a satisfying and safe sexual life and using their reproductive abilities.

Sexual and reproductive health and rights are essential for the health and survival of people, economic development and prosperity. In the United Nations 2030 Sustainable Development Goals, the third article named "Health and Quality Life" includes the targets covering reproductive health and sexual health. Some of these goals are; universal access to sexual and reproductive health services, creation of national education and information strategies for reproductive health, preventing sexually transmitted infections (STIs), access to information about family planning, and reducing maternal and neonatal mortality. People can lead a complete healthy and quality life only when these goals are achieved.

It is observed that the knowledge of men and women about general reproductive health and the organs and functions of the female and male reproductive systems is significantly lacking. In addition to these, it has been reported that they have insufficient knowledge on other issues such as sexual health, STIs and family planning methods. There are studies showing that lack of knowledge brings about reproductive health problems in young individuals. Problems such as exposure to STIs, early pregnancy, and risky sexual behaviors arise due to lack of information. Since all these health problems can cause permanent damage, the individual's future reproductive health is also at risk. However, it is possible to come across studies showing that reproductive health education is a tool to prevent these adverse health conditions. In a study conducted with university students, even if students' basic sexual education knowledge levels were good; It has been reported that there is a positive relationship between receiving sexual education and protective sexual behaviors, knowledge, motivation and skills. At the same time, it has been reported in many studies that believing in sexual myths, which are considered as false beliefs and have no scientific value, is more common in students with high levels of knowledge. While sexual myths cause behavioral changes with believed mistakes, sexual dysfunctions, decrease in sexual satisfaction and negative attitude towards contraceptive methods can also be brought about. Considering that people who know more about sexually transmitted HIV/AIDS have a low rate of believing in myths, an important reproductive health problem such as STI should be considered to be related to myths.

In this context, training on reproductive health and sexual health is important. Preparation and implementation of trainings on reproductive and sexual health by health professionals; It is important as it is known that young people have access to conflicting or incorrect information from various sources. Therefore, health professionals should be involved in these training processes. While planning the trainings, many platforms can be used, and nowadays, web-based trainings increase their importance with the introduction of the internet in all areas of our lives. The biggest advantages of web-based education are that it can be accessed anytime, anywhere and by anyone. In various studies conducted with university students, it is seen that web-based education increases the level of knowledge and is effective in behavior change.

In this period when technological education emerged, many instructional design models developed were used in web-based education. Among these models, the most widely used ADDIE model. ADDIE is a model that provides a systematic and comprehensive definition and implementation of design principles. The web-based training in the research will be given based on the ADDIE Model approach. Basic elements of the instructional design process in the model; It is in the form of Analysis, Design, Development, Implementation and Evaluation. The use of a model in web-designed education ensures that the educational content is prepared according to the needs, the training steps are not skipped and systematic.

In the literature review and web researches, a web-based education was not encountered in national and international publications where university students could reach the correct and scientific information about reproductive health. In this context, the investigators believe that web-based education to be provided with the ADDIE Model approach will reduce the sexual myths and risky behaviors that young people believe.

This study was planned to examine the effect of web-based reproductive health education given to university students on belief in sexual myths and risky behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year undergraduate / associate degree student
* Not taking any anatomy or women's health classes
* Volunteering to participate in research
* Being in the age range of 18-24

Exclusion Criteria:

* Voluntarily leaving the research
* Not attending the trainings given in the experimental group

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Baseline (To both groups before the intervention)
  This form, which was prepared by the researchers by scanning the literature, in order to describe the sociodemographic and reproductive health information of the students participating in the study, and the platforms / individuals from which this information was obtained, consists of 20 questions.
Sexual Myths Scale | Change in believing sexual myths at Baseline and 5 weeks of education)
  It is a scale developed to describe sexual myths scale by Gölbaşı et al. in 2016. The scale consists of 8 sub-dimensions and 28 items that allow the multidimensional evaluation of sexual myths.
  Sub Dimensions and Item Numbers; Sexual orientation: 1-5. Articles, Gender: 6-11. Substances, Age and sexuality: 12-15. Substances, Sexual behavior: 16-18. Substances, Masturbation: 19-20. Sexual violence: 21-24. Substances, Sexual intercourse: 25-26. Substances, Sexual Satisfaction: 27-28. Substances. Each item of the scale is evaluated on a 5-point: "Never agree" = 1, "Disagree" = 2, "Undecided" = 3, "Partially Agree" = 4, "Strongly Agree" = 5. The total score for the scale is obtained by adding the scores given to each item. The minimum score obtained from the scale is 28 and the maximum score is 140. The scale does not have a cut-off point. The higher the score, the higher the sexual myths.
Information and Risky Behavior Form Specific to Reproductive Health Education | Change in risky behavior at Baseline and 5 weeks of education)
  It is a form consisting of 47 questions created after the literature review. Contains; male and female anatomy and physiology, regulation of fertility, sexually transmitted infections and risky behaviors related to these issues. The items in the form consist of true and false statements that evaluate students' knowledge and attitudes about risky behaviors in the educational content. The questions in each item will be answered as "True, False, No Idea". The questions in the form will be submitted for expert opinion. A pre-test will be conducted to detect the presence of incomprehensible expressions. The score of the form will be calculated by giving 1 point to each correct answer and the highest score will be 47.

CONTACTS AND LOCATIONS:
Locations (1):
- Güzin Ünlü, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aggarwal, A. K., & Bento, R. (2002). Web-based education. In Web-based instructional learning (pp. 59-77). IGI Global.
- [Background] Ancheta R, Hynes C, Shrier LA. Reproductive health education and sexual risk among high-risk female adolescents and young adults. J Pediatr Adolesc Gynecol. 2005 Apr;18(2):105-11. doi: 10.1016/j.jpag.2005.01.005. PMID 15897107
- [Background] Apay, S. E., Akpınar, R. B., & Arslan, S. (2013). Öğrencilerin cinsel mitlerinin incelenmesi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 16(2), 96-102.
- [Background] Apay, S. E., Nagorska, M., Akpınar, R. B., Celik, A. S., & Binkowska-Bury, M. (2013). Student comparison of sexual myths: two-country case. Sexuality and Disability, 31(3), 249-262.
- [Background] Aronowitz T, Lambert CA, Davidoff S. The role of rape myth acceptance in the social norms regarding sexual behavior among college students. J Community Health Nurs. 2012;29(3):173-82. doi: 10.1080/07370016.2012.697852. PMID 22857406
- [Background] Aygin, D., Açıl, H., Yaman, Ö., & Çelik Yılmaz, A. (2017). Üniversitede okuyan kadın öğrencilerin cinsel mitler ile ilgili görüşleri. Androloji Bülteni, 19(2), 44-49.
- [Background] Baghaie, R., Rasouli, D., Rahmani, A., Mohammadpour, Y., & Jafarizade, H. (2012). Effect of web-based education on cardiac disrhythmia learning in nursing student of Urmia University of Medical Sciences. Iranian Journal of Medical Education, 12(4), 240-248.
- [Background] Çetin, Ö., & Aslan, E. (2019) Adölesanlarda Sık Görülen Jinekolojik Sorunlar. Sağlık Bilimlerinde İleri Araştırmalar Dergisi, (2), 33-43.
- [Background] Duan YP, Wienert J, Hu C, Si GY, Lippke S. Web-Based Intervention for Physical Activity and Fruit and Vegetable Intake Among Chinese University Students: A Randomized Controlled Trial. J Med Internet Res. 2017 Apr 10;19(4):e106. doi: 10.2196/jmir.7152. PMID 28396306
- [Background] Gölbaşı, Z. (2005). Adölesan Dönem Üreme Sağlığı Sorunları Ve Etkileyen Faktörler. Anadolu Hemşirelik Ve Sağlık Bilimleri Dergisi, 8(1), 100-108.
- [Background] İpek, İ., Sözcü, Ö. F., & Ziatdinov, R. (2013). Birleştirilmiş E-Öğrenme Tasarımı Modeli ve Hızlı Öğretim Tasarımı Stratejileri. Akademik Bilişim Konferansı, Akdeniz Üniversitesi Hukuk Fakültesi Antalya-Türkiye (http://ab. org. tr/ab13/bildiri/).
- [Background] Kalembo, F. W., Zgambo, M., & Yukai, D. (2013). Effective adolescent sexual and reproductive health education programs in sub-Saharan Africa. Californian Journal of Health Promotion, 11(2), 32-42.
- [Background] Kukulu, K., Gürsoy, E., & Sözer, G. A. (2009). Turkish university students' beliefs in sexual myths. Sexuality and Disability, 27(1), 49-59.
- [Background] Michie L, Cameron ST, Glasier A, Wellings K, Loudon J. Myths and misconceptions about intrauterine contraception among women seeking termination of pregnancy. J Fam Plann Reprod Health Care. 2014 Jan;40(1):36-40. doi: 10.1136/jfprhc-2012-100497. Epub 2013 May 24. PMID 23709608
- [Background] Moradi, A., Salimi, M., Esfarjani, S. V., & Haghighizadeh, M. H. (2017). Effect of Web-based education on knowledge and preventive behaviors of Iron Deficiency Anemia among high school girls. Journal of Clinical and Analytical Medicine, 1, 445.
- [Background] Özerbaş, M. A., & Kaya, A. B. (2017). Öğretim Tasarımı Çalışmalarının İçerik Analizi: ADDIE Modeli Örneklemi. Journal Of Turkish Educational Sciences, 15(1).
- [Background] Reis, M., Ramiro, L., de Matos, M. G., & Diniz, J. A. (2011). The effects of sex education in promoting sexual and reproductive health in Portuguese university students. Procedia-Social and Behavioral Sciences, 29, 477-485.
- [Background] Solikhah, S. N. (2015). Knowledge and behaviour about adolescent reproductive health in Yogyakarta, Indonesia. International Journal of Public Health, 4(4), 326-331.
- [Background] Starrs AM, Ezeh AC, Barker G, Basu A, Bertrand JT, Blum R, Coll-Seck AM, Grover A, Laski L, Roa M, Sathar ZA, Say L, Serour GI, Singh S, Stenberg K, Temmerman M, Biddlecom A, Popinchalk A, Summers C, Ashford LS. Accelerate progress-sexual and reproductive health and rights for all: report of the Guttmacher-Lancet Commission. Lancet. 2018 Jun 30;391(10140):2642-2692. doi: 10.1016/S0140-6736(18)30293-9. Epub 2018 May 9. No abstract available. PMID 29753597
- [Background] Teitelman AM, Bohinski JM, Boente A. The social context of sexual health and sexual risk for urban adolescent girls in the United States. Issues Ment Health Nurs. 2009 Jul;30(7):460-9. doi: 10.1080/01612840802641735. PMID 19544131
- [Background] Tenkorang EY. Myths and misconceptions about HIV transmission in Ghana: what are the drivers? Cult Health Sex. 2013;15(3):296-310. doi: 10.1080/13691058.2012.752107. Epub 2012 Dec 14. PMID 23240740
- [Background] Terzioglu F, Kok G, Guvenc G, Ozdemir F, Gonenc IM, Hicyilmaz BD, Sezer NY. Sexual and Reproductive Health Education Needs, Gender Roles Attitudes and Acceptance of Couple Violence According to Engaged Men and Women. Community Ment Health J. 2018 Apr;54(3):354-360. doi: 10.1007/s10597-017-0227-3. Epub 2018 Jan 15. PMID 29335810
- [Background] United Nations (UN). (2015). The 2030 Agenda For Sustainable Development. access link: https://sustainabledevelopment.un.org/content/documents/21252030%20Agenda%20for%20Sustainable%20Development%20web.pdf Access Date:14.06.2020
- [Background] Wang, S. K., & Hsu, H. Y. (2008, November). Using ADDIE model to design Second Life activities for online learners. In E-Learn: World Conference on E-Learning in Corporate, Government, Healthcare, and Higher Education (pp. 2045-2050). Association for the Advancement of Computing in Education (AACE).
- [Background] Wong LP. An exploration of knowledge, attitudes and behaviours of young multiethnic Muslim-majority society in Malaysia in relation to reproductive and premarital sexual practices. BMC Public Health. 2012 Oct 11;12:865. doi: 10.1186/1471-2458-12-865. PMID 23057505
- [Background] World Health Organization (WHO) (2008). Integrating poverty and gender into health programmes: a sourcebook for health professionals: module on sexual and reproductive health. Access Lİnk: https://apps.who.int/iris/bitstream/handle/10665/206996/9789290613893_eng.pdf?sequence=1&isAllowed=y Access Date: 14.06.2020